CLINICAL TRIAL: NCT02798406
Title: A Phase II, Multi-center, Open-label Study of a Conditionally Replicative Adenovirus (DNX-2401) With Pembrolizumab (KEYTRUDA®) for Recurrent Glioblastoma or Gliosarcoma (CAPTIVE/KEYNOTE-192)
Brief Title: Combination Adenovirus + Pembrolizumab to Trigger Immune Virus Effects
Acronym: CAPTIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DNAtrix, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2401BT-002P
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Brain Cancer; Brain Neoplasm; Glioma; Glioblastoma; Gliosarcoma; Malignant Brain Tumor; Neoplasm, Neuroepithelial; Neuroectodermal Tumors; Neoplasm by Histologic Type; Neoplasm, Nerve Tissue; Nervous System Diseases
Keywords: brain; Central Nervous System (CNS) diseases; Central Nervous System (CNS) neoplasms; CNS; conditionally replicative adenovirus; DNX-2401; pembrolizumab; KEYTRUDA; MK-3475; SCH 900475; lambrolizumab; neoplasm, germ cell and embryonal; neoplasm, granular and epithelial; Alcyone; Alcyone Lifesciences; AMC; cannula; MEMS cannula; DNX-2401 + pembrolizumab; Delta-24; Delta-24-RGD; Checkpoint inhibitor; anti-PD1/PD-L1; immunotherapy; monoclonal antibody; KEYNOTE-192
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Gliosarcoma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms, Nerve Tissue; Nervous System Diseases; Disease; Neoplasms | interventions — Oncolytic Virotherapy; pembrolizumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DNX-2401 + pembrolizumab (Experimental): Intratumoral dose (1.0 mL) of DNX-2401 followed 7-9 days later by intravenous pembrolizumab, 200 mg, given every three weeks through 105 weeks (2 yrs.) or until progressive disease or unacceptable toxicity.
  Interventions: Biological: DNX-2401; Biological: pembrolizumab

INTERVENTIONS:
Biological: DNX-2401 — On Day 0, following brain tumor biopsy and confirmation of recurrent tumor, a single injection of DNX-2401 is administered directly into the brain tumor.
  Other Names: Oncolytic virus; Genetically-modified adenovirus; Delta-24; Delta-24-RGD
Biological: pembrolizumab — Sequential intravenous administration every three weeks beginning 7-9 days after Day 0/DNX-2401
  Other Names: KEYTRUDA; lambrolizumab; MK-3475; SCH 900475; Checkpoint inhibitor; monoclonal antibody; anti-PD1/PD-L1

SUMMARY:
Glioblastoma (GBM) and gliosarcoma (GS) are the most common and aggressive forms of malignant brain tumor in adults and can be resistant to conventional therapies. The purpose of this Phase II study is to evaluate how well a recurrent glioblastoma or gliosarcoma tumor responds to one injection of DNX-2401, a genetically modified oncolytic adenovirus, when delivered directly into the tumor followed by the administration of intravenous pembrolizumab (an immune checkpoint inhibitor) given every 3 weeks for up to 2 years or until disease progression.

Funding Source-FDA OOPD

DETAILED DESCRIPTION:
In the initial phase of the study, up to 12 evaluable subjects will be enrolled in 3 dose cohorts to determine the best dose of DNX-2401, as follows:

* Cohort 1: Single dose DNX-2401 (5e8 vp) delivered intratumorally by cannula, followed by intravenous pembrolizumab every 3 weeks (Q3W)
* Cohort 2: Single dose DNX-2401(5e9 vp) delivered intratumorally by cannula, followed by intravenous pembrolizumab every 3 weeks (Q3W)
* Cohort 3: Single dose DNX-2401 (5e10 vp) delivered intratumorally by cannula, followed by intravenous pembrolizumab every 3 weeks (Q3W)

Following the initial phase, up to 36 additional subjects diagnosed with recurrent glioblastoma or gliosarcoma will be enrolled to receive a single of DNX-2401 determined in the initial phase administered intratumorally followed by intravenous pembrolizumab every 3 weeks.

All subjects will return to the clinic for study follow-up visits at regular intervals for safety monitoring, MRI scans and other assessments, for up to 2 years or until disease progression. All subjects will be followed closely for safety and survival.

ELIGIBILITY:
Inclusion Criteria:

* A single glioblastoma or gliosarcoma tumor with histopathological confirmation for first or presenting second recurrence of glioblastoma or gliosarcoma at the time of consent
* Gross total or partial tumor resection is not possible or not planned
* A single measurable tumor that is at least 10.0 mm longest diameter (LDi) X 10.0 mm shortest diameter (SDi) and this tumor does not exceed 40.0 mm in LDi or SDi on Screening MRI
* Tumor recurrence or progression documented after previously failing surgical resection, chemotherapy or radiation
* Karnofsky performance status ≥ 70 %
* Prior anti-tumor therapies must have been completed within time periods specified in the protocol prior to DNX-2401 injection and toxic side effects must be mild, if present
* Demonstrate adequate organ function via specified laboratory test results

Exclusion Criteria:

* Multiple (≥ 2) separate enhancing tumors
* Tumor location on both sides of the brain and/or involvement that would present the risk of injecting DNX-2401 into the ventricles of the brain
* Tumor location in the brain stem
* Requires or, based upon history, may require treatment with high-dose systemic corticosteroids within 2 weeks of the start of intravenous pembrolizumab infusions and within 2 weeks following the first infusion of pembrolizumab
* Uncontrolled blood-sugar levels defined as HbA1c > 7%
* Previous treatment with any checkpoint inhibitor such as anti-PD1 or PD-L1 agents including pembrolizumab (KEYTRUDA) or any other checkpoint inhibitor(s) (e.g., ipilimumab, nivolumab, etc.)
* History of (non-infectious) or current active pneumonitis that required steroids and/or a history of interstitial lung disease
* Prior gene transfer therapy or prior therapy with a cytolytic virus of any type
* Brain tumor that is not measurable on MRI or persons who are unable to have MRIs
* Pregnant or nursing females

Note: Other protocol-defined inclusion and exclusion criteria may apply as outlined in the relevant protocol version

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3.5 years
  Interval tumor size reduction as measured from periodic MRI

SECONDARY OUTCOMES:
Overall survival (OS) | 3.5 years
  Months alive following treatment as measured during periodic study visits
Time to tumor response | 3.5 years
  Months to response following treatment as measured during periodic MRIs
Duration of response | 3.5 years
  Months of sustained response as measured during periodic study visits

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gady, BS, Study Director — DNAtrix, Inc.
Locations (15):
- United States (14):
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Minnesota Neurosurgery, Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill-Cornell Medicine New York-Presbyterian, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University James Cancer Center, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Texas Oncology Austin-Midtown, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Plan to share aggregate data at completion of study

REFERENCES:
- [Derived] Nassiri F, Patil V, Yefet LS, Singh O, Liu J, Dang RMA, Yamaguchi TN, Daras M, Cloughesy TF, Colman H, Kumthekar PU, Chen CC, Aiken R, Groves MD, Ong SS, Ramakrishna R, Vogelbaum MA, Khagi S, Kaley T, Melear JM, Peereboom DM, Rodriguez A, Yankelevich M, Nair SG, Puduvalli VK, Aldape K, Gao A, Lopez-Janeiro A, de Andrea CE, Alonso MM, Boutros P, Robbins J, Mason WP, Sonabend AM, Stupp R, Fueyo J, Gomez-Manzano C, Lang FF, Zadeh G. Oncolytic DNX-2401 virotherapy plus pembrolizumab in recurrent glioblastoma: a phase 1/2 trial. Nat Med. 2023 Jun;29(6):1370-1378. doi: 10.1038/s41591-023-02347-y. Epub 2023 May 15. PMID 37188783